CLINICAL TRIAL: NCT04453449
Title: A Prospective Study Investigating the Effect of Midazolam Sedation on Diagnostic Lumbar Medial Branch Blocks
Brief Title: The Effect of Midazolam Sedation on Diagnostic Medial Branch Blocks
Acronym: MBB
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Katherine Nowak, Research Manager, Henry Ford Health System
Other Study IDs: 14010
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Lumbar Spine Spondylosis; Anxiety Generalized
Keywords: midazolam; sedation; diagnostic lumbar medial branch block; radiofrequency thermocoagulation
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Midazolam

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- No sedation: Patients who will undergo the diagnostic lumbar medial branch blocks without sedation (control group).
- Sedation: Patients who will undergo the diagnostic lumbar medial branch blocks with midazolam sedation (treatment group).
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — Midazolam given as a sedative during diagnostic lumbar medial branch block
  Other Names: sedation
  Groups: Sedation

SUMMARY:
This prospective observational study aims to investigate the effect of midazolam sedation on the diagnostic validity of diagnostic lumbar medial branch block in patients diagnosed with lumbar spondylosis without myelopathy.

DETAILED DESCRIPTION:
This prospective observational study aims to investigate the effects of midazolam sedation on the diagnostic validity of lumbar medial branch blocks in patients diagnosed with lumbar spondylosis without myelopathy. Patients typically receive two subsequent diagnostic blocks prior RFTC, to ensure that the correct location has been targeted. When patients achieve at least 80% pain relief after both diagnostic blocks, this is considered a positive result and they can proceed to receive RFTC. If patients have positive diagnostic blocks but their RFTC is not successful, this is considered a false positive diagnostic result. This study will determine 1) if a higher number of sedated patients proceed to radiofrequency thermocoagulation (RFTC) than non-sedated patients, and 2) if there are a higher number of false positive results in sedated patients. The hypothesis is that the use of midazolam sedation will increase the number of patients who perceive to have pain relief from their diagnostic block results, resulting in more patients proceeding to RFTC, and that there will be a higher number of false positive results in sedated patients. The primary outcome measure is the number of sedated versus non-sedated patients that have positive block results. A positive result will be calculated by having at least one NRS score that is at least 80% lower than their baseline NRS score in the 8 hours following lumbar MBB. The secondary outcome will be the number of false positive blocks in sedated versus non-sedated patients. After patients achieve 80% relief after each of the two diagnostic lumbar medial branch blocks and proceeds with lumbar RFTC, we will then collect NRS scores 24 hours after both diagnostic Lumbar MBB, and 4 weeks and at 8 weeks after the lumbar RFTC. If a patient has not received at least 50% reduction from their baseline NRS score by 8 weeks, this will be considered a false positive. A 7-point Patient Global Impression of Change (PGIC) score 8 hours after each Lumbar MBB will also be collected, and at 4 weeks and 8 weeks after the lumbar RFTC, and any adverse effects patients experience. In addition, Oswestry Disability Index (ODI) will be collected at 4 and 8 weeks after lumbar RFTC. The results of this study will help guide the use of sedation when performing diagnostic blocks on patients with lumbar spondylosis, in order to reduce the number of false positive blocks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at least 18 years of age
* History of axial low back pain for at least 3 months
* Indication for bilateral lumbar medial branch block (L3, L4, L5 medial branch nerves)
* Diagnosis of Lumbar Spondylosis without Myelopathy >4/10 pain on a 0-10 numerical rating scale (NRS)

Exclusion Criteria:

* Low back pain with radiculopathy symptoms (this is a diagnosis of sciatica and treatment is not with lumbar medial branch block)
* Uncontrolled major depression or other mental health issues causing instability
* Pregnant or lactating women
* <18 years old
* History of adverse reaction to either midazolam, lidocaine, or bupivacaine
* Focal neurological deficits, cognitive impairments, or memory issues
* Non-English speaking
* Hearing impaired that are unable to understand verbal instructions
* Active Infection
* On Anticoagulation or Antiplatelet Therapy
* History of Clotting Disorder
* Previous Lumbar Medial Branch Block and/or Lumbar Radiofrequency Ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with Lumbar Spondylosis without Myelopathy at either of five study locations (HFMC - Ford Rd, HFMC Main, HFMC West Bloomfield, HFMC Pierson, HFMC - Jackson) from June 1st, 2020 - June 1st, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Number of positive blocks | 8 hours post diagnostic block
  The number of positive diagnostic lumbar medial branch blocks (defined by at least 80% pain relief) in patients who receive midazolam sedation during their diagnostic blocks will be compared to patients who do not receive sedation.

SECONDARY OUTCOMES:
Number of false positive blocks | 2.5-3 months
  The number of false positive diagnostic lumbar medial branch blocks (defined by at least 80% pain relief in the two diagnostic blocks, and then less than 80% pain relief following the subsequent radiofrequency thermocoagulation treatment) in patients who receive midazolam sedation during their diagnostic blocks will be compared to patients who do not receive sedation.

OTHER OUTCOMES:
Patient Global Impression of Change-7 (PGIC-7) scores | 24 hours post diagnostic block; 4 and 8 weeks after radiofrequency thermocoagulation
  The PGIC-7 scores of patients who received sedation will be compared to those who did not receive sedation during their diagnostic lumbar medial branch block.
Oswestry Disability Index (ODI) scores | 4 and 8 weeks after radiofrequency thermocoagulation
  The ODI scores of patients who received sedation will be compared to those who did not receive sedation during their diagnostic lumbar medial branch block.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Derived] Patel N, Nowak K, Vaidyanathan A, Milad H, Adlaka K, Rubino C, Vasquez ET, Nerusu L, Rahavard B, Fayed M, Forrest P, Money S, Dwivedi S, Zador L, Haddad R, Khaja D, Sibai N, Aiyer R. The Effect of Sedation on Diagnostic Lumbar Medial Branch Blocks for Facetogenic Low Back Pain: An Observational Study. Pain Physician. 2024 May;27(4):E407-E418. PMID 38805536